CLINICAL TRIAL: NCT00002671
Title: PHASE II STUDY OF 9-20-S-AMINO-CAMPTOTHECIN (9-AC) AS SECOND LINE THERAPY IN ADVANCED OVARIAN CARCINOMA
Brief Title: Aminocamptothecin in Treating Patients With Recurrent or Unresectable Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000064290; NYU-9501; E-9501; NCI-T95-0001D
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2006-05

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Drug: aminocamptothecin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of aminocamptothecin in treating patients with recurrent or unresectable epithelial ovarian cancer that has been previously treated with platinum-based chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate in patients with advanced, recurrent, or inoperable ovarian epithelial cancer treated with aminocamptothecin as second-line therapy. II. Determine the toxic effects of this regimen in these patients. III. Correlate the topoisomerase-I levels with response in patients with accessible tumors treated with this regimen.

OUTLINE: Patients are stratified according to disease (measurable vs nonmeasurable). (The measurable disease stratum closed to accrual effective 08/1998.) Patients receive aminocamptothecin IV continuously on days 1-3. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) receive 4 additional courses past CR. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients (30 per stratum) will be accrued for this study within approximately 15 months. (The measurable disease stratum closed to accrual effective 08/1998.)

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced, recurrent, or inoperable ovarian epithelial cancer Previously treated with 1 platinum-containing chemotherapy regimen Bidimensionally measurable or reproducibly measurable disease in 2 dimensions on CT scan (The measurable disease stratum closed to accrual effective 08/1998) OR Evaluable but radiographically nonmeasurable disease with CA-125 more than 50 units/mL on 2 measurements at least 1 week apart

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT and SGPT no greater than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No myocardial infarction, congestive heart failure, or other significant cardiac disease within the past 6 months No uncontrolled hypertension Other: No significant active infection (e.g., pneumonia, peritonitis, or wound abscess) No uncontrolled metabolic disease (e.g., diabetes mellitus or hypothyroidism) No asthma (even if controlled with medication) No other serious concurrent illness No dementia or altered mental status that would preclude informed consent No other malignancy except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: See Disease Characteristics No more than 1 prior chemotherapy regimen No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: See Disease Characteristics Other: At least 4 weeks since prior investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-12; Primary Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (6):
- United States (6):
  - Riverview Medical Center, Red Bank, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York

REFERENCES:
- [Result] Hochster H, Plimack ER, Runowicz CD, Speyer J, Wallach RC, Sorich J, Mandeli J, Wadler S, Wright J, Muggia FM. Biweekly 72-hour 9-aminocamptothecin infusion as second-line therapy for ovarian carcinoma: phase II study of the New York Gynecologic Oncology Group and the Eastern Cooperative Oncology Group. J Clin Oncol. 2004 Jan 1;22(1):120-6. doi: 10.1200/JCO.2004.03.016. PMID 14701774
- [Result] Speyer JL, Hochster H, Runowicz C, et al.: Phase II study of 72 hr 9-amino-camptothecin (9AC) infusion in second-line therapy of ovarian cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A1401, 363a, 1999.